CLINICAL TRIAL: NCT01956682
Title: Hypoallergenic Infant Formula Containing Starch and the Probiotic: Effect on Gastric Emptying
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Bari (Other)
Responsible Party: Principal Investigator, Flavia Indrio, M.D., University of Bari
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: University of Bari
Record Dates: First submitted 2013-09-18; First posted 2013-10-08 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2015-03

CONDITIONS: Regurgitation, Gastric
MeSH Terms: conditions — Laryngopharyngeal Reflux | interventions — Starch

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Infant formula (Active Comparator): HA formula + starch + L. reuteri
  Interventions: Dietary Supplement: HA formula + starch + L. reuteri
- Standard Formula (Placebo Comparator): Standard Infant Formula

INTERVENTIONS:
Dietary Supplement: HA formula + starch + L. reuteri
  Arms: Infant formula

SUMMARY:
The primary objective of this trial is to show that an hypoallergenic infant starter formula containing starch and the probiotic L. reuteri decreases the severity of regurgitation/spitting-up in infants presenting regurgitation/spitting-up , and who have taken it for 4 weeks, in comparison with a standard infant starter formula.

DETAILED DESCRIPTION:
The primary objective of this trial is to show that the test formula (HA formula + starch + L. reuteri) decreases the severity (frequency + volume) of regurgitation/spitting-up in infants and ultrasound gastric emptying time, compared to a classical infant starter formula.

ELIGIBILITY:
Inclusion Criteria:

* Full term infant (37 weeks ≤ gestation ≤ 42 weeks)
* Age of infant between 5 days and 5 months
* NGA
* Infant exclusively formula-fed at enrollment
* Presenting regurgitation/spitting-up according to the parents' perception
* Vandenplas score of at least 2 and maximum 5
* Having obtained the subject's legal representative's written informed consent

Exclusion Criteria:

* Previous antireflux treatment
* Previous consumption of AR infant formula or external thickener
* Previous consumption of a formula with L. reuteri
* Cow's milk allergy symptoms according to medical decision
* Congenital illness or malformation that may affect growth
* Significant pre-natal and/or post-natal disease
* Newborn whose parents / caregivers cannot be expected to comply with study procedures
* Newborn currently participating or having participated in another clinical trial during the last 4 weeks prior to the beginning of this study.

Ages: 5 Days to 5 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 132 (Actual)
Dates: Start 2014-10; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Regurgitation | four weeks of treatment
  The primary outcome is the difference in the proportions of improved subjects at four weeks of treatment between the treatment and control groups.

SECONDARY OUTCOMES:
Growth | Four weeks of treatment
  To assess whether the groups have comparable growth
Regurgitation score | Four weeks treatment
  To assess the severity of regurgitation/spitting-up To assess the frequency of regurgitation/spitting-up To assess the volume of regurgitation/spitting-up
Gastric empty rate | Four week treatment
  To compare the ultrasound gastric empty rate
Digestive tolerance | Four weeks treatment
  To assess the infants' digestive tolerance
Stool frequency | Four weeks treatment
  To assess stool frequency
compliance | four weeks intervention
  To assess the subject's compliance to product consumption.
Financial and non-financial burden | Four week treatment
  To measure family financial and non-financial burden related with the regurgitation

CONTACTS AND LOCATIONS:
Overall Officials: Flavia Indrio, MD, Principal Investigator — University of Bari
Locations (1):
- Ospedale Pediatrico Giovanni XXIII, Bari, BA, Italy